CLINICAL TRIAL: NCT04235413
Title: Impact of Real-Time Incentives on Fruit and Vegetable Purchases and Diet
Brief Title: Fruits and Vegetables Incentives Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 833359
Record Dates: First submitted 2020-01-08; First posted 2020-01-21 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Fruit and Vegetable Intake; Healthy Diet
Keywords: nutrition; health disparities; food purchases
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-Time Incentives Group (Experimental): Each participant will be randomized using a blocking procedure (SNAP participant or not). The intervention will last 6 months and consist of receiving real-time financial incentives at the point of purchase for eligible fruits and vegetables purchases.
  Interventions: Behavioral: Real-Time Incentives Group
- Control Group (No Intervention): No intervention administered. Each participant will be randomized using a blocking procedure (SNAP participant or not).

INTERVENTIONS:
Behavioral: Real-Time Incentives Group — The use of a novel computer program with a mobile phone interface to provide real-time financial incentives at the point of purchase for discounts on fruit and vegetables in low-income families. This intervention will be applied to subjects randomized to the intervention arm. They will receive 50% off eligible fruits and vegetable products at the point of purchase, up to $10 a week for 6 months. Maximum amount they can receive is $260 in discounts over the 6 month period.
  Arms: Real-Time Incentives Group

SUMMARY:
The goal of this study is to evaluate the effectiveness of financial incentives delivered in real-time at point of purchase, on low-income consumers' purchase of fruits and vegetables, fruits and vegetables consumption, diet quality, and weight/BMI. The study will test real-time incentives compared to a no-incentive control condition.

DETAILED DESCRIPTION:
To address diet quality disparities in low-income families, policy makers and health experts recommend strategies such as financial incentives to promote consumption of fruits and vegetables. Real-time incentives for purchasing fruits and vegetables are promising strategies to improve families' diets and health.

The aims of the study are:

1. To test the effects of financial incentives, delivered in real-time at the point of purchase, on low-income consumer purchases of fruits and vegetables
2. To evaluate the impact of real-time financial incentives compared to a control condition on FV consumption among adults and their children ,shopping habits, home food environments, diet quality, and weight/BMI
3. To adapt mobile platform technology to provide regular feedback to participants to motivate use of the incentive program to increase purchases and consumption of fruits and vegetables
4. To evaluate participant satisfaction with real-time healthy food choice incentives technology in both SNAP participants and income-eligible non-SNAP participants
5. To assess the acceptability and ease of use of real-time healthy food choice incentives technology among retails supermarket managers and staff in low-income neighborhoods.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Speak English
* Do most of their food shopping at a participating supermarket
* Receive or are eligible to receive SNAP benefits
* Have a child in the household between the ages of 2-17
* Have a working smartphone
* Be the main household shopper

Exclusion Criteria:

* Participants will be excluded if the primary shopper and/or any children in the family have major medical or dental conditions that would prevent them from eating fruits and vegetables, or if they have a serious neurological disorder, dementia, or psychiatric condition that interferes with understanding study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Self-reported fruits and vegetables (FV) purchase data | up to 8 months
  Participants will be asked if they increased, maintained, or decreased their purchases of canned, frozen, and fresh FV in the previous months.
Intake of fruits and vegetables (FV) per day | Baseline, 6 months, 8 months
  FV consumption intake will be assessed using the Dietary Screener Questionnaire from NHANES (National Healthy and Examination Survey) 2009-2010.

SECONDARY OUTCOMES:
Total mean of fruits and vegetables expenditures/purchases and incentives earned | up to 8 months
  Solutran analytics, our partner that will be delivering the incentives, will be providing weekly data on FV expenditures/purchases and incentives earned (in dollars). The total mean of FV expenditures/purchases and incentives earned will be computed.
Dietary changes for each adult participant and one child in their household | Baseline, 6 months, 8 months
  High sugar/fat food and sugary beverage intake will be assessed using the Dietary Screener Questionnaire from NHANES (National Healthy and Examination Survey) 2009-2010.
Changes in dietary habits and food environments | Baseline, 6 months, 8 months
  Surveys will ask about perceived availability, cost and quality of FV at stores, the home food environment (both healthy and unhealthy foods), shopping habits and where they shop, FV practices for children in the home, and FV preparation and consumption patterns. Part of the survey is a modified version of the NEMS-P (Nutrition Environment Measures Survey- Perceived).
Changes in BMI | Baseline, 6 months, 8 months
  Self-reported weight and height (inches) will be collected at each time point via self-report. Using weight and height values collected, BMI, BMI categories, and BMI z-scores (for children) will be computed for each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Glanz, PhD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided